CLINICAL TRIAL: NCT04961528
Title: ACid Tranexamic or Terlipressin for Initial Emergency Treatment of Mild to seVere hEmoptysis: a Randomized Trial.
Acronym: ACTIVE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP200043; 2020-005931-58 (EudraCT Number); PHRC-19-0412 (Other Grant/Funding Number: French ministry of health)
Record Dates: First submitted 2021-07-05; First posted 2021-07-14 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Hemoptysis
Keywords: terlipressin; tranexamic acid
MeSH Terms: conditions — Hemoptysis | interventions — Tranexamic Acid; Terlipressin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Terlipressin (Experimental): Dosage: 1 mg /5 ml Pharmaceutical form: solution for infusion Posology: 1 mg /8 hours Treatment duration: 3 days
  Method and route of administration: inhalation using the same jet nebulizers (INT'AIR Medical RN 300) in all Investigating centers
  Interventions: Drug: Terlipressin
- Tranexamic Acid (Experimental): Dosage : 500 mg /5 ml Pharmaceutical form: solution for infusion Posology (and adjustments based on toxicity) : 500 mg/ 8 hours Treatment duration: 3 days
  Method and route of administration: inhalation using the same jet nebulizers (INT'AIR Medical RN 300) in all Investigating centers.
  Interventions: Drug: Tranexamic Acid 500 MG
- Normal Saline Placebo (Placebo Comparator): Dose : normal saline solution (NaCl 0.9%) Pharmaceutical form : solution for infusion Posology : 5ml / 8 hours Treatment duration: 3 days
  Method and route of administration: inhalation using the same jet nebulizers (INT'AIR Medical RN 300) in all Investigating centers.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid 500 MG — Jet nebulization (a device connected by tubing to compressed air or oxygen to flow at high velocity through a liquid medicine to turn it into an aerosol, which is then inhaled by the patient).
  The nebulization lasts 10 minutes. Posology: 500 mg x 3/day (= 500 mg / 8 hours) Treatments duration: 3 days
  Arms: Tranexamic Acid
Drug: Terlipressin — Jet nebulization (a device connected by tubing to compressed air or oxygen to flow at high velocity through a liquid medicine to turn it into an aerosol, which is then inhaled by the patient).
  The nebulization lasts 10 minutes. Posology: 1 mg x 3/day (= 1 mg / 8 hours) Treatments duration: 3 days
  Arms: Terlipressin
Drug: Placebo — Jet nebulization (a device connected by tubing to compressed air or oxygen to flow at high velocity through a liquid medicine to turn it into an aerosol, which is then inhaled by the patient).
  The nebulization lasts 10 minutes. Posology: 5ml x 3/day (= 5 ml / 8 hours) Treatments duration: 3 days.
  Other Names: Normal saline placebo
  Arms: Normal Saline Placebo

SUMMARY:
The study aims is to verify the hypothetize that inhaled Tranexamic Acid (TXA) or Terlipressin (TER) will be associated with an increase in the rapid control of hemoptysis without side-effects.

This randomized double-blind multicenter triple arm trial compares the administration of TXA to TER to placebo in patients with mild to severe hemoptysis.

DETAILED DESCRIPTION:
In over 90% of cases, hemoptysis is due to a bronchial or non-bronchial systemic arterial mechanism.

Embolization of Bronchial Arteries (EBA) is the main specific treatment but is not easily available. Medical treatment for hemoptysis is not evidence-based.

For this study, the investigators will dispense trial drugs using inhalation route which has not been evaluated in mild to severe hemoptysis in previous trials. In addition, as opposed to previous trials, the investigators will assess the safety of trials drugs during hospital stay.

Acid tranexamic (TXA), an antifibrinolytic drug, reduces bleeding in uterine and traumatic haemorrhage by blocking the action of plasmin on fibrin. Intravenous terlipressin (TER), a vasoconstrictor, contributes to control digestive haemorrhage but presents many contraindication when administrated by intravenous route.

The investigator hypothetize that inhaled antifibrinolytic (TXA) or vasoconstrictor (TER) will be associated with an increase in the rapid control of hemoptysis without side-effects.

Patients will be randomized into 3 groups:

* Active treatment 1: Tranexamic Acid 500 mg three times a day (every 8 hours) for 5 days.
* Active treatment 2: Terlipressin 1 mg three times a day (every 8 hours) for 5 days.
* Placebo: normal saline nebulization three times a day (every 8 hours) for 5 days.

Using a hierarchical analysis, the comparison between TXA and TER will be tested once superiority on efficacy of both inhaled TXA and TER vs placebo is demonstrated. The above secondary objectives will then be assessed for the comparison of TXA versus TER.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years, under 90 years
* Mild to severe hemoptysis that has been going on for less than 7 days
* Total expectorate blood ranging from 50 ml to 200 ml
* Admission in emergency department or ICU for less than 12 hours
* Social security affiliation
* Signed informed consent
* For child-bearing aged women, efficient contraception includes oral oestrogen- progestin, oral progestin, progestin implants and all types of intrauterine devices

Exclusion Criteria:

* Need for mechanical ventilation
* Cystic fibrosis
* Pregnancy or breast feeding
* Contraindication for contrast agents injection (renal failure with creatinin clearance < 30mL/min, know allergy to contrast agents injection)
* Known hypersensitivity to TXA or TER or one of its excipients
* Know previous cardiac arrhythmia (atrial fibrillation, atrial flutter..)
* Contraindication to TXA (including renal failure with creatinin clearance < 30mL/min) or TER therapy :

  * acute myocardial infarction in the 6 past months,
  * intrathecal injection in the 3 past months,
  * seizure in the past 3 months
* Participation in another interventional study or being in the exclusion period at the end of a previous study.
* Patient under tutorship or / guardianship, and incapable to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2022-03-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with complete or partial resolution of hemoptysis without the use of any interventional procedure. | 3 days
  Efficacy of inhaled tranexamic acid and inhaled terlipressin versus placebo (normal saline) in immediate control of mild to severe hemoptysis within the first 3 days of hospitalization.
  A complete resolution of hemoptysis is defined by absence of recurrence within 3 days; partial resolution is defined as hemoptysis recurrence < 50 ml within the first 3 days

SECONDARY OUTCOMES:
Rate of complete resolution of hemoptysis within 3 days, as previously defined | 3 days
  Complete resolution of hemoptysis, as previously defined
Rate of partial resolution of hemoptysis defined as recurrence < 50 ml | 3 days
  Partial resolution of hemoptysis, as previously defined
Rate of patients with total volume of hemoptysis < 200 ml | 3 days
  Total volume of hemoptysis < 200 ml
Rate of patients who need an endovascular treatment (bronchial arterial endovascular embolization) | 3 days
  Need of invasive procedure such as bronchial arterial endovascular embolization
Time between hospital admission and bronchial arterial endovascular embolization | 3 days
  Time between hospital admission and endovascular treatment
Rate of patients who need a mechanical ventilation | 3 days
  Need of invasive procedure such as mechanical ventilation,
Rate of specific adverse events | 3 days
  Specific Adverse Events (AE) : acute myocardial ischemia, symptomatic venous thromboembolism, hyponatremia (<130 mmol/L), bronchospasm (defined by the need of short-acting bronchodilatator).
Rate of in-hospital mortality | 30 days
Rate of patients with hemoptysis recurrence | 30 days
Death rate | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Planquette, MD, PhD, Study Chair — AP-HP, Hôpital Européen Georges Pompidou, Paris
Locations (1):
- AP-HP, Hôpital Européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Teams wishing obtain IPD must meet the sponsor and PI team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasability and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).